CLINICAL TRIAL: NCT05118334
Title: An Open Label, Multicenter, Phase Ib Study Evaluating IBI310 (Anti-CTLA-4) in Combination With Sintilimab in Patients With Advanced, Recurrent or Metastatic Non-small-cell Lung Cancer (NSCLC)
Brief Title: IBI310 (Anti-CTLA-4) in Combination With Sintilimab in Patients With Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310H201
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: NSCLC (Non-small-cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IBI310 (anti-CTLA-4) 1mg/kg(Q3W until progressive disease)in combination with Sintilimab (Experimental): The test group will be treated with IBI310 1mg/kg IV, Q3W+ Sintilimab 200 mg IV, Q3W until progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: IBI310
- IBI310 (anti-CTLA-4) 1mg/kg(Q3W*4cycles)in combination with Sintilimab (Experimental): The test group will be treated with IBI310 1mg/kg IV, Q3W+ Sintilimab 200 mg IV, Q3W*4cycles,and then Sintilimab 200 mg IV, Q3W single until progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: IBI310
- IBI310 (anti-CTLA-4) 1mg/kg(Q6W)in combination with Sintilimab (Experimental): The test group will be treated with IBI310 1mg/kg IV, Q6W+ Sintilimab 200 mg IV, Q3Wuntil progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: IBI310
- IBI310 (anti-CTLA-4) 0.5mg/kg in combination with Sintilimab (Experimental): The test group will be treated with IBI310 0.5mg/kg IV, Q3W+ Sintilimab 200 mg IV, Q3W until progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: IBI310

INTERVENTIONS:
Drug: Sintilimab — (IBI310 1mg/kg IV, Q3W+ Sintilimab 200 mg IV, Q3W)until progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
Drug: IBI310 — (IBI310 1mg/kg IV, Q3W+ Sintilimab 200 mg IV, Q3W) until progressive disease,intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.

SUMMARY:
This is an open label, multicenter, phase Ib study evaluating IBI310 (anti-CTLA-4) in combination with Sintilimab in patients with advanced, recurrent or metastatic non-small-cell lung cancer (NSCLC)

ELIGIBILITY:
Eligibility Criteria:

1. Aged ≥18 years;
2. ECOG 0 ~ 1;
3. Histologically /cytologically confirmed R/M NSCLC;
4. Adequate organ and bone marrow function;
5. Expected survival ≥12 weeks;
6. Female subjects of childbearing age or male patients whose sex partners are women of childbearing age should take effective contraceptive measures throughout the treatment period and within 6 months after the last administration;
7. Subjects who sign the written informed consent form, and can abide by the visits and related procedures specified in the protocol.
8. At least 1 measurable lesion according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST V1.1).

Exclusion Criteria:

1. Had tumors other than NSCLC within the past 5 years.
2. Had allogeneic organ or stem cell transplantation.
3. The presence of uncontrolled life-threatening illness
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Patients who have used large doses of glucocorticoids, anti-cancer monoclonal antibodies, and other immunosuppressive agents within 4 weeks.
6. HIV positive.
7. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
8. Severe, uncontrolled medical conditions and infections.
9. At the same time using other test drugs or in other clinical trials.
10. Refusal or inability to sign informed consent to participate in the trial.
11. Other treatment contraindications.
12. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.
13. Hepatitis B surface antigen (HBsAg) positive and HBVDNA ≥1000cps/ml.
14. Patients with positive HCV antibody test results can only be included in the study when the polymerase chain reaction of HCV RNA is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to 2 years
  Investigator evaluated ORR per RECIST V1.1
Treatment Emergent Adverse Event (TEAE) | Up to 2 years
  Incidence and severity of treatment-emergent: which is evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v5.0) grade;
Severe Adverse Event (SAE) | Up to 2 years
  Incidence and severity of treatment-emergent: which is evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v5.0) grade;

SECONDARY OUTCOMES:
DOR | Up to 2 years
  Defined as the time from the first documented objective response to the first documented progressive disease or death of any cause, whichever occurs first;
Progression Free Survival (PFS) | Up to 2 years
  Defined as the time from randomization to the first documented progressive disease or death of any cause, whichever occurs first;
Overall Survival (OS) | Up to 2 years
  Defined as the time from randomization to death of any cause in subjects without receiving any immunotherapy outside the study protocol for first-line treatment of advanced NSCLC
Disease Control Rate (DCR) | Up to 2 years
  Defined as the proportion of patients whose best response is CR, PR, and stable disease (SD) non-CR/non-PD
Time to Response (TTR) | Up to 2 years
  Defined as the time from randomization to the first documented and confirmed objective response (CR or PR)
HRQoL | Up to 2 years
  According to EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Chen X, Yao J, Long J, Mao Y, Wu D, Zang A, Zhao J, Liu Z, Meng R, Chen Y, Luo Y, Guo Q, Li L, Cui J. A phase Ib study evaluating the safety and efficacy of IBI310 plus sintilimab in patients with advanced non-small-cell lung cancer who have progressed after anti-PD-1/L1 therapy. Cancer Med. 2024 Feb;13(3):e6855. doi: 10.1002/cam4.6855. Epub 2024 Jan 12. PMID 38214075